CLINICAL TRIAL: NCT03378999
Title: A Proof of Concept Study to Demonstrate a Cholesterol-lowering Benefit of Oven-dried Rhodospirillum Rubrum
Brief Title: Rhodospirillum Rubrum and Cholesterol
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: ezCOL B.V. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: METC17-3-026
Record Dates: First submitted 2017-12-06; First posted 2017-12-20 (Actual); Last update posted 2019-05-24 (Actual); Status verified 2019-03

CONDITIONS: Cholesterol Metabolism

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control (Placebo Comparator): Placebo capsules containing microcrystalline cellulose
  Interventions: Dietary Supplement: Control
- Rhodospirillum rubrum 0.25 gram/day (Experimental): Capsules containing oven-dried Rhodospirillum rubrum, 0.25 gram/day
  Interventions: Dietary Supplement: Rhodospirillum rubrum
- Rhodospirillum rubrum 0.5 gram/day (Experimental): Capsules containing oven-dried Rhodospirillum rubrum, 0.5 gram/day
  Interventions: Dietary Supplement: Rhodospirillum rubrum
- Rhodospirillum rubrum 1.0 gram/day (Experimental): Capsules containing oven-dried Rhodospirillum rubrum, 1.0 gram/day
  Interventions: Dietary Supplement: Rhodospirillum rubrum

INTERVENTIONS:
Dietary Supplement: Rhodospirillum rubrum — Capsules containing oven-dried Rhodospirillum rubrum
  Arms: Rhodospirillum rubrum 0.25 gram/day; Rhodospirillum rubrum 0.5 gram/day; Rhodospirillum rubrum 1.0 gram/day
Dietary Supplement: Control — Capsules containing microcrystalline cellulose
  Arms: Control

SUMMARY:
The primary objective of the study is to examine for the first time the LDL cholesterol lowering effect of oven-dried Rhodospirillum rubrum in humans.

DETAILED DESCRIPTION:
Objectives:

Secondary objectives are to investigate the effects on other CVD risk parameters: total cholesterol, triacylglycerol, HDL-C, glucose and blood pressure. Safety will be monitored by measurements of markers for liver, kidney and heart function.

Study design:

The study is a 4-weeks randomized, double-blind placebo-controlled trial with a parallel design using 3 doses oven-dried Rhodospirillum rubrum. Prior to and after the intervention period, a 2-week run-in and run-out period takes place, during which all subjects will consume placebo capsules.

Study population:

Eighty (N=80) healthy men with a slightly elevated fasting serum total cholesterol concentration (between 5.0-8.0 mmol/l) will complete the study.

Intervention:

During the intervention period of 4 weeks, men will receive either placebo or capsules containing 0.25 gr, 0.5 gr or 1.0 gr oven-dried Rhodospirillum rubrum per day.

ELIGIBILITY:
Inclusion Criteria:

* Minimum 80 kg body weight;
* Serum total cholesterol between 5.0 - 8.0 mmol/L (further testing is recommended for excessive hyperlipidemia [serum total cholesterol ≥ 8.0 mmol/L] according to the Standard for cardiovascular risk management of the Dutch general practitioners community [NHG]);
* Serum triacylglycerol concentrations < 4.5 mmol/L;
* No signs of liver and/or kidney dysfunction;
* No diabetic patients;
* No familial hypercholesterolemia;
* No abuse of drugs;
* Not more than 4 alcoholic consumption per day with a maximum of 21 per week;
* Stable body weight (weight gain or loss < 3 kg in the past three months);
* No use of medication known to treat blood pressure, lipid or glucose metabolism;
* No use of an investigational product within another biomedical intervention trial within the previous 1-month;
* No severe medical conditions that might interfere with the study, such as epilepsy, asthma, kidney failure or renal insufficiency, chronic obstructive pulmonary disease, inflammatory bowel diseases, auto inflammatory diseases and rheumatoid arthritis;
* No active cardiovascular disease like congestive heart failure or cardiovascular event, such as an acute myocardial infarction or cerebrovascular accident;
* Willingness to give up being a blood donor from 8 weeks before the start of the study, during the study and for 4 weeks after completion of the study;
* No difficult venipuncture as evidenced during the screening visit;
* Willing to comply to study protocol during study;
* Informed consent signed.

Exclusion Criteria:

* Serum total cholesterol < 5.0 mmol/L or ≥ 8.0 mmol/L;
* Serum triacylglycerol concentrations ≥ 4.5 mmol/L;
* Signs of liver and/or kidney dysfunction;
* Diabetic patients;
* Familial hypercholesterolemia;
* Abuse of drugs;
* More than 4 alcoholic consumptions per day or 21 per week;
* Unstable body weight (weight gain or loss > 3 kg in the past three months);
* Use medication known to treat blood pressure, lipid or glucose metabolism;
* Use of an investigational product within another biomedical intervention trial within the previous 1-month;
* Severe medical conditions that might interfere with the study, such as epilepsy, asthma, kidney failure or renal insufficiency, chronic obstructive pulmonary disease, inflammatory bowel diseases, auto inflammatory diseases and rheumatoid arthritis;
* Active cardiovascular disease like congestive heart failure or cardiovascular event, such as an acute myocardial infarction or cerebrovascular accident;
* Not willing to give up being a blood donor from 8 weeks before the start of the study, during the study or for 4 weeks after completion of the study;
* Not or difficult to venipuncture as evidenced during the screening visit;
* Use of over-the-counter and prescribed medication or supplements, which may interfere with study measurements to be judged by the principal investigator;
* Use of oral antibiotics in 40 days or less prior to the start of the study;
* Blood donation in the past 3 months before the start of the study;
* Not willing to comply to study protocol during study or sign informed consent.

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2018-06-14 (Actual); Primary Completion 2019-05-10 (Actual); Study Completion 2019-05-10 (Actual)

PRIMARY OUTCOMES:
LDL cholesterol concentrations | Change from baseline LDL cholesterol concentrations at 4 weeks
  Fasting LDL cholesterol concentrations will be determined in blood samples using the Friedewald equation

SECONDARY OUTCOMES:
Markers for fasting lipid metabolism | Change from baseline concentrations at 4 weeks
  Markers for fasting lipid metabolism include serum total cholesterol (mmol/L), HDL cholesterol (mmol/L), and triacylglycerol concentrations (mmol/L).
Glucose concentrations | Change from baseline concentrations at 4 weeks
  Fasting plasma glucose concentrations will determined in blood samples
Blood pressure | Change from baseline blood pressure at 4 weeks
  Systolic and diastolic blood pressure
C-reactive protein | hs-CRP will be will be measured at day 0, day 14, day 25 and day 28 of the intervention period
  Concentrations of hs-CRP will be determined in blood samples
Markers for liver function | These markers will be measured at day 0, day 14, day 25 and day 28 of the intervention period
  Markers for liver function include ALAT, ASAT and yGT (U/L). This panel of markers will be assessed to monitor liver function.
Markers for kidney function | These markers will be measured at day 0, day 14, day 25 and day 28 of the intervention period
  Markers for kidney function include creatinine
Markers for heart function (NT-ProBNP) | These markers will be measured at day 0, day 14, day 25 and day 28 of the intervention period
  Markers for heart function include NT-ProBNP. This panel of markers will be assessed to monitor heart function.
Markers for heart function (vWF) | These markers will be measured at day 0, day 14, day 25 and day 28 of the intervention period
  Markers for heart function include vWF. This panel of markers will be assessed to monitor heart function.
Markers for heart function (Troponin-T) | These markers will be measured at day 0, day 14, day 25 and day 28 of the intervention period
  Markers for heart function include Troponin-T. This panel of markers will be assessed to monitor heart function.

CONTACTS AND LOCATIONS:
Overall Officials: Jogchum Plat, MSc, Principal Investigator — Maastricht University Medical Center
Locations (1):
- Maastricht University Medical Center, Maastricht, Limburg, Netherlands